CLINICAL TRIAL: NCT07003100
Title: A Prospective, US-Based Study Assessing Mogamulizumab-Associated Rash in Patients Diagnosed With Mycosis Fungoides or Sézary Syndrome and Treated With Standard of Care Mogamulizumab
Brief Title: A Prospective, US-based Study Assessing Mogamulizumab-associated Rash in Patients Diagnosed With Mycosis Fungoides or Sezary Syndrome and Treated With Standard of Care Mogamulizumab
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22233; NCI-2024-01011 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22233 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-06-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Mycosis Fungoides; Recurrent Sezary Syndrome; Refractory Mycosis Fungoides; Refractory Sezary Syndrome; Stage IB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIA Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage III Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IV Mycosis Fungoides and Sezary Syndrome AJCC v8
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete questionnaires, have photographs of their skin taken, and undergo blood sample collection and skin biopsies on study. Patients' medical records are also reviewed.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to assess mogamulizumab-associated rash in patients diagnosed with mycosis fungoides or sezary syndrome and treated with standard of care mogamulizumab. One of the most common side effects of mogamulizumab is a rash, currently named mogamulizumab-associated rash (MAR) which can look like MF or SS. However, mogamulizumab-associated rash (MAR) does not indicate failure of mogamulizumab, and may be a sign that the drug is working. If not properly evaluated, mogamulizumab-associated rash (MAR) could be misinterpreted as worsening of mycosis fungoides/sezary syndrome, which could lead doctors to recommend stopping mogamulizumab treatment early. The information learned by doing this research study may help tell the difference between mogamulizumab-associated rash (MAR) (sometimes also called "drug eruption") and worsening of the disease. It may also help to uncover information about the cause of mogamulizumab-associated rash (MAR).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the incidence of mogamulizumab-associated rash (MAR) and its association with overall response in patients with cutaneous T-cell lymphoma (CTCL); mycosis fungoides [MF] and sezary syndrome [SS] subtypes) treated with mogamulizumab.

OUTLINE: This is an observational study.

Patients complete questionnaires, have photographs of their skin taken, and undergo blood sample collection and skin biopsies on study. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* * Adult patients (>= 18 years of age) diagnosed with relapsed/refractory Mycosis Fungoides (MF) stage IB, IIA, IIB, III and IV or Sezary Syndrome(SS), and selected by their treating physician to receive single agent mogamulizumab (newly initiated)

  * Signed informed consent
  * Willing to undergo baseline biopsy and during treatment to evaluate for Mogamulizumab-Associated Rash (MAR) if clinically indicated
  * Willing to provide blood sample at baseline, and if applicable, at onset of Mogamulizumab-Associated Rash (MAR)

Exclusion Criteria:

* * Other concomitant systemic and skin directed Cutaneous T-cell Lymphoma (CTCL) regimens except for topical steroids

  * Prior treatment with mogamulizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with relapsed/refractory Mycosis Fungoides (MF) stage IB, IIA, IIB, III and IV or Sezary Syndrome(SS), and selected by their treating physician to receive single agent mogamulizumab (newly initiated).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Binary incidence of mogamulizumab-associated rash (MAR) | Up to 3 years
  Will be estimated as a binomial proportion along with the 95% exact binomial confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Querfeld, Principal Investigator — City of Hope Medical Center
Locations (10):
- United States (10):
  - City of Hope Medical Center, Duarte, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington